CLINICAL TRIAL: NCT01263392
Title: A Comparison of the Incidence of Symptomatic Urinary Tract Infections in Children With Spina Bifida Using Hydrophilic or Non-hydrophilic Polyvinyl Chloride Catheters for Clean Intermittent Catheterization: a Randomized Cross Over Trial
Brief Title: Comparing Urinary Tract Infections in Children With Spina Bifida Using Two Types of Catheters for Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Speedi 10
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-03

CONDITIONS: Neurogenic Bladder; Spina Bifida
Keywords: Neurogenic bladder; Spina bifida; Intermittent catheterization; Urinary tract infections
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Dysraphism; Urinary Tract Infections | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyvinyl Chloride Catheter (Active Comparator): Re-use clean polyvinyl chloride catheters for intermittent catheterization of children with spina bifida.
  Interventions: Device: Intermittent catheterization
- Hydrophilic catheter (Active Comparator): Use hydrophilic catheters (Speedicath) for intermittent catheterization of children with spina bifida.
  Interventions: Device: Intermittent catheterization

INTERVENTIONS:
Device: Intermittent catheterization — Subjects will use each type of catheter for 6 months and will report weekly in a diary on urinary tract infections (UTIs), urine dip for haematuria & leukocytes, antibiotic use, and days missed school; and will answer a Satisfaction questionnaire at the end of each 6 month arm.
  Other Names: Polyvinyl Chloride; Hydrophillic - Coloplast Speedicath catheter

SUMMARY:
The primary aim of this study was to determine if using the SpeediCath hydrophilic catheter would reduce the incidence of symptomatic urinary tract infections (UTI)in children with spina bifida who perform clean intermittent catheterization for bladder management. The hypothesis was that the incidence of symptomatic urinary tract infections would be significantly reduced (by 25%) in users of the SpeediCath hydrophilic catheter when compared to users of a reused polyvinyl chloride (PVC) catheter. Subjects were randomly assigned to either starting the study with PVC catheter for 6 months followed by the hydrophilic catheter for 6 months or visa versa. Each subject kept a weekly diary recording urinary tract infections symptoms, hematuria determined by urine dipstick, physician visits, days of missed school and other activities. At the end of each 6 months subjects completed a questionnaire recording their comfort and satisfaction in using the PVC or hydrophilic coated catheter. 70 subjects were randomized and 46 had complete data. There were no differences in febrile UTI, antibiotic use, healthcare visits or school days missed. The incidence of self reported UTI was lower in the PVC group than the hydrophilic group. 40% of subjects indicated that the hydrophilic coated catheter was slippery and difficult to handle compared to 10% for the PVC catheter. However overall satisfaction was no different between products. The study results are consistent with the current Cochrane Review that there is a lack of evidence to state that the incidence of UTI is affected by multiuse or hydrophilic catheter use.

DETAILED DESCRIPTION:
Intermittent catheterisation (IC) is accepted management for maintaining bladder and renal health in individuals with incomplete bladder emptying. Two common products are available for IC: polyvinyl chloride (PVC) and single use hydrophilic coated PVC. In 2004 the UK spent around £33 million on hydrophilic catheters compared to £3 million for PVC catheters. Proposed advantages of the lubricated hydrophilic catheter over PVC catheters are:

1. lower incidence of symptomatic urinary tract infections (UTI) and
2. lower incidence of urethral irritation, trauma and urethral strictures from repeated IC.

Complications and UTIs are costly to the individual and the system but despite over 25 RCTs on the topic, there remains a lack of evidence indicating superiority of one product over another in community dwelling IC users.

Purpose: To compare the incidence of symptomatic UTI in children with spina bifida using single use hydrophilic (SpeediCath™) or PVC catheters for IC. Secondary aims: compare differences in weekly urinalysis for blood and leukocytes; physician visits, antibiotic use, days missed of school or activities; subject and care provider satisfaction with study catheter products.

Study Design, materials and methods: Randomised crossover two arm trial at four Western Canada paediatric sites: each arm was 24 weeks of single use hydrophilic or PVC catheters cleaned with soap and water (standard of care). Symptomatic UTI defined as positive leukocytes plus > 1 fever, flank pain, increased incontinence, malaise, cloudy or odorous urine requiring antibiotic treatment. Randomisation was determined at the study centre using a computer generated list into random block sizes of 8. Subject assignments were placed in opaque envelopes and sealed. After consent was obtained the local research assistant contacted the site technician who opened the envelope and gave the assignment. Sample size: With power of 80%, an expected difference of 25% between treatment and control and α 0.05, the total sample size needed was 97 subjects, using methods for correlated binary data and repeated measures. All data was entered by an impartial technician. It was not possible to blind subjects to product. Data were analyzed using a Mixed Within-Subjects Between-Subjects Analysis of Variance where the group was defined by the catheter type on which the trial began. SPSS version 20 was used for all analyses.

Inclusion Criteria: Child with spina bifida living in the community who either self IC or received IC by a consistent person; child/parent/caregiver able to read and understand English. Exclusion criteria: Urethral deformities (i.e. stricture, false passage); antibiotic prophylaxis; allergy to PVC product; diabetes mellitus; history of bladder pathology (i.e. tumours, calculus); surgical history of augmentation (cystoplasty, continent diversion).

Results: 70 subjects were randomized; 46 had complete data over 48 weeks; 24 dropouts: hydrophilic catheter too slippery (15%); refused PVC arm because they preferred hydrophilic catheter (5%); booked for continent diversion (4%), other (8%). Mean age 10.6 (SD 6.2), 21 males and 25 females. All performed IC > 3/day: 52% self and 48% parents/ caregivers; PVC catheters were used at least 5 times. Mean total weeks of self-reported UTI was 3.6 (SD 4.7) in the hydrophilic group vs. 2.3 (SD 3.3) in the PVC group (p= <.001) but no statistical differences in weeks of febrile UTI, antibiotic use, visits to physicians, days missed from school, or microscopic haematuria (urine dip). There was a trend to fewer weeks of positive leukocytes in the hydrophilic group (Table 1).

There were no statistically significant differences in Convenience or Comfort. Ease of Handling was significantly different with 40% disliking the hydrophilic product compared to 10% for the PVC product. Fewer participants answered "yes" to "would you continue using the product" (hydrophilic vs. the PVC 65% vs. 90% respectively). However, overall satisfaction was no different between products (Table 2).

Interpretation of Results:

The study was underpowered despite major attempts at recruitment. However the findings are clinically relevant. The hydrophilic catheter was more difficult to handle and therefore less likely to be continued than the PVC multiuse product. Participants who overcame the handling issues found the product excellent. Incidence febrile UTI or of antibiotic treated UTI did not appear to be affected by single use vs. multiuse products.

Conclusions: A hydrophilic catheter does not appear to reduce febrile UTI or antibiotic use in community dwelling children using CIC. Attrition was high based on participants' lack of adjustment to the hydrophilic product and to study fatigue. The study results are consistent with the existing Cochrane Review: there is a lack of evidence to state the incidence of UTI is affected by multiuse or hydrophilic catheter use. Large multicentre trials are strongly recommended.

Table 1: Mean number of weeks (of 24) with Symptoms Hydrophilic Single Use PVC multiuse N Mean N Mean Leucocytes 50 8.46 52 10.10 Fever 50 .04 49 .06 Other Symptoms ( w no Fever) 50 3.50 49 2.22 Hematuria 50 2.64 52 3.15 Antibiotics 50 .80 49 .55 Days Missed Activities 50 .40 52 .13 Note: all comparisons p>0.05

Table 2: Overall satisfaction with catheter products Hydrophilic Single Use PVC multiuse N % Acceptable N % Acceptable Convenience 49 81.6 48 81.3 p>0.05 Comfort 48 87.5 47 95.7 p>0.05 Ease of handling 49 59.2 48 95.8 p<0.05 Would you continue to use? 49 57.1 48 91.7 p<0.05 Overall satisfaction 48 72.9 48 87.5 p>0.05

ELIGIBILITY:
Inclusion Criteria:

* Healthy Child with spina bifida who requires clean intermittent catheterization (CIC) for ongoing bladder management.
* Child either self catheterizes or receives catheterization by a consistent person.
* Child/parent/caregiver able to read and understand English in order to consent to participation in the study and to respond to verbal questions about the experience and satisfaction with the catheter.

Exclusion Criteria:

* Urethral deformities (i.e. stricture, false passage)
* Antibiotic prophylaxis
* Allergy to PVC product
* Diabetes Mellitus
* Unwilling to reuse catheters
* History of bladder pathology (ie. tumours, calculus)
* Surgical history of augmentation (cystoplasty, continent diversion)

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2007-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Symptomatic urinary tract infection (UTI) | 6 months and 6 months at crossover
  Symptomatic urinary tract infection (UTI) as per CDC definitions

SECONDARY OUTCOMES:
Subject satisfaction | 6 months and 6 months at cross over
  Comparative data between polyvinyl chloride (PVC) and hydrophilic catheter on convenience, comfort, ease of handling, continuing to use, and overall satisfaction recorded on validated Satisfaction Questionnaire by subject

OTHER OUTCOMES:
urinalysis (urine dipstick) | 6 months and 6 months at crossover points
  urinalysis --- presence of leukocytes, haematuria as measured by subject and recorded in weekly diary
Antibiotic use for any reason | 6 months and 6 months at cross over points
  Antibiotic use recorded by subject
Physician or healthcare provider visits | 6 months and 6 months at crossover points
  physician visits for any reason
Effect on daily activities | 6 months and 6 months at crossover
  days missed of school or activities as recorded by subject in weekly diary

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Moore, PhD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, Winnipeg, Manitoba